CLINICAL TRIAL: NCT00338663
Title: The Effect of Knee Immobilization on Postoperative Pain Following an Anterior Cruciate Ligament (ACL) Reconstruction: A Randomized Clinical Trial
Brief Title: A Study on Knee Immobilization and Pain Levels After an Anterior Cruciate Ligament (ACL) Reconstruction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeMark Health Research Group (Other)
Collaborators: LifeMark Health (Other); Calgary Orthopaedic Research and Education Fund (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: E-20041
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: anterior cruciate ligament reconstruction; knee immobilization; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: knee immobilization splint

SUMMARY:
The purpose of the study is to determine if there is difference in immediate postoperative pain levels (48 hours) between patients who wear a knee immobilizer splint compared to patients who do not wear a knee immobilizer splint after an anterior cruciate ligament reconstruction surgery.

DETAILED DESCRIPTION:
This study will attempt to evaluate the efficacy of knee immobilization on patient postoperative pain levels following an ACL reconstruction. There is a lack of consensus in the area of postoperative knee bracing/immobilization. A survey of Canadian surgeons indicates that the primary reason for postoperative knee immobilization is to reduce pain. To the investigators' knowledge, there are no studies comparing the use of immediate (0-48 hours) postoperative knee immobilization versus no immobilization and pain control in this patient population.

ELIGIBILITY:
Inclusion Criteria:

- Clinical: Patients' aged 18-40, ACL deficiency as determined by MRI or physical exam (positive lachmann and pivot shift tests) resulting in giving way episodes (acute or chronic) unresponsive to non-operative management and therefore requiring primary ACL reconstruction.

- Arthroscopic: Concomitant meniscal resection.

Exclusion Criteria:

- Clinical: Previous surgery on either knee (not including a diagnostic arthroscopy arthroscopy or simple partial meniscectomy,) Concomitant lower extremity fracture, Ipsilateral collateral ligament injury within past 3 months, Time from ACL injury less than 6 weeks, Allergy/intolerance to Tylenol 3 with codeine and to Percocet, Third Party or Medical Legal.

- Radiological: Skeletal immaturity (open growth plates).

- Arthroscopic/surgical: Concomitant posterior cruciate ligament or collateral ligament repairs, Osteochondral lesions requiring microfracture, Meniscal repair, Patients not having both their semitendinosus and gracilis harvested.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88
Dates: Start 2006-05; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Patient self-assessed pain levels using an unmarked zero to one hundred mm visual analog scale (VAS) at forty eight hours postoperative.

SECONDARY OUTCOMES:
Patient self-assessed pain levels using an unmarked zero to one hundred mm visual analog scale (VAS) at seven and fourteen days postoperative.
Analgesic type and time taken will be self reported by the patient at each VAS entry.
Range of motion including both flexion and extension will be assessed at fourteen days postoperative by the surgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie A Hiemstra, MD, PhD, Principal Investigator — LifeMark Health Research Group
Locations (2):
- Canada (2):
  - Banff Sport Medicine Clinic, Banff, Alberta
  - Lindsay Park Sports Injury Clinic, Calgary, Alberta